CLINICAL TRIAL: NCT00710216
Title: Randomized, Open-Label, Phase IV Trial in Nucleus(t)id-Naive Patients With Chronic Hepatitis B to Examine the Effect of Telbivudine Compared to Lamivudine on the Early Dynamics and Kinetics of Viral Suppression (Early-Viral-Dynamics Study)
Brief Title: Comparison of Telbivudine Versus Lamivudine on the Early Dynamics and Kinetics of Viral Suppression in Chronic Hepatitis B
Acronym: EVD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdraw
Sponsor: University of Ulm (Other)
Collaborators: Novartis (Industry)
Responsible Party: PD Dr. med. Nektarios Dikopoulos, Universitätsklinikum Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVD-001
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Hepatitis B, Chronic
Keywords: Viral kinetics; Viral dynamics; Telbivudine; Lamivudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; lipoarabinomannan; Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Lamivudine
- B (Experimental)
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Lamivudine — 100 mg/day
  Other Names: Zeffix; Epivir; LAM; 134678-17-4; J05AF05; 73339
  Arms: A
Drug: Telbivudine — 600 mg/day
  Other Names: Sebivo; Tyzeka; L-dT; 3424-98-4; J05AF11; 159269
  Arms: B

SUMMARY:
This study examines the effect of telbivudine compared to lamivudine on the early viral kinetics in patients with chronic hepatitis B. The virus Kinetics is measured by the viral load (HBV-DNA) reduction in the serum during the first 12 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented compensated HBeAg-positive or negative chronic hepatitis B
* Increased viral load with a concentration of serum HBV-DNA of at least 10^4 copies/ml
* Proof of inflammatory activity in the liver: ALT ≥ 2 x ULN or histological evidence of inflammatory activity ≥ level I or fibrosis of ≥ I degrees (according to the Desmet classification)
* Negative urine pregnancy test with fertile women
* Willingness to use a recognized method of contraception
* Able to comply with study regimen and provide written informed consent

Exclusion Criteria:

* Current or previous antiviral treatment of chronic hepatitis B with Nucleus(t)id analoga
* Known hypersensitivity to lamivudine or telbivudine or any of the other components of the preparations
* Pregnant or breastfeeding women or women
* Simultaneous participation in other clinical trials or in the past three months
* Co-infected with HCV, HDV, HIV
* Other non HBV-related chronic liver disease: Autoimmune hepatitis, primary biliary cirrhosis, Hemochromatosis, alpha-1 antitrypsin deficiency, alcoholic hepatitis
* Evidence of hepatocellular carcinoma (alpha-fetoprotein levels> 100 ng/ml)
* Active drug use, including an excessive alcohol consumption during the last 6 months before participating in the clinical trial
* Use of systemic treatment with anti-neoplastic or immunomodulatory medication within the last 6 months before participating in the clinical trial and during the duration of the clinical examination
* Lack of willingness or inability to consent in writing
* Concurrent condition likely to preclude compliance with schedule of evaluations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
Decrease in viral load after 2 weeks of therapy measured in serum HBV-DNA concentration (Copies/ml or IU/ml). | 2 weeks

SECONDARY OUTCOMES:
Course of the viral load (serum HBV-DNA) during the first 12 weeks of therapy | 12 weeks
Influence of HBeAg status to the decrease in viral load | 12 weeks
Influence of HBV genotype to the decrease in viral load | 12 weeks
Change in ALT and AST levels from Baseline to Week 12 | 12 weeks
Development of viral resistance and treatment failure during the study and subsequent course of observation | 6 month
Safety assessed by adverse events and laboratory values | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Nektarios Dikopoulos, MD, Principal Investigator — University Hospital Ulm
Locations (1):
- University Hospital Ulm, Ulm, Germany

REFERENCES:
- See also: University Hospital Ulm — http://www.uniklinik-ulm.de/